CLINICAL TRIAL: NCT04142502
Title: Comparison of the Effects of Dexmedetomidine and Propofol on the Cardiovascular Autonomic Nervous System During Spinal Anesthesia: Pilot Study
Brief Title: Comparison of the Effects of Dexmedetomidine and Propofol on the Cardiovascular Autonomic Nervous System During Spinal Anesthesia
Acronym: ANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Ilsung Pharmaceuticals CO.,LTD. (Unknown)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MED-INT-19-350
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Spinal Anesthesia; Autonomic Nervous System
Keywords: spinal anesthesia; autonomic nervous system; dexmedetomidine; propofol
MeSH Terms: interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Propofol group: propofol infusion as sedation drug Dexmedetomidine group: dexmedetomidine infusion as sedation drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Active Comparator): Using propofol as a sedation drug Infusion rate control Effect site concentration 0.3~1.0 mg/ml using target concentration infusion Bispectral index 60~80
  Interventions: Drug: Propofol
- Dexmedetomidine group (Active Comparator): Using dexmedetomidine as a sedation drug First 10 minutes 1.0 mcg/kg loading After 10 minutes 0.3-1.0 mcg/kg/hr maintenance Bispectral index 60~80
  Interventions: Drug: Dexmedetomidin

INTERVENTIONS:
Drug: Propofol — Propofol as a sedation drug
  Other Names: FRESofol MCT inj 1% 500mg/50ml, Fresenium Kabi
  Arms: Propofol group
Drug: Dexmedetomidin — Dexmedetomidine as a sedation drug
  Other Names: Medex inj, 200mcg/2ml, ILSUNG
  Arms: Dexmedetomidine group

SUMMARY:
Spinal anesthesia induces bradycardia and hypotnesion, because itself decreases parasympathetic activity and increases sympathetic activity. These imbalance of autonomic nervous system can be measured by heart rate variability. Propofol and dexmedetomidine, which are used for sedation during spinal anesthesia, also affect autonomic nervous system, but the exact effects are not well known. The purpose of this study is measuring the effects of propofol or dexmedetomidine on autonomic nervous system in spinal anesthesia.

DETAILED DESCRIPTION:
Spinal anesthesia induces bradycardia and hypotnesion, because itself decreases parasympathetic activity and increases sympathetic activity. These imbalance of autonomic nervous system can be measured by heart rate variability. Propofol and dexmedetomidine, which are used for sedation during spinal anesthesia, also affect autonomic nervous system but the exact effects are not well known. Moreoever, the effect of spinal anesthesia combined with sedation agent on autonomic nervous system has not been evaluated. The purpose of this study is measuring the effects of propofol or dexmedetomidine on autonomic nervous system in spinal anesthesia. The current study is prospective randomized pilot study. Patients are assigned to propofol group and dexmedetomidine group. Using electrocardiaogram analysis, the change of autonomic nervous system will be measured from preoperative to end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 20~60 years old
* Scheduled lower extremity surgery under spinal anesthesia

Exclusion Criteria:

* Arryhthmia
* Uncooperative patients
* Diabetes
* On medication: beta blocker, psychiatric medicine
* Thyroid function abnormality

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Serial heart rate variability | 40 minutes (before entering the operating room ~ 20 minutes after starting sedation
  Serial change of frequency domain results from EKG RR interval Baseline: before entering the operating room T0: Preinduction T1: 10 minutes after spinal anesthesia T2: 10 minutes after starting sedation T3: 20 minutes after starting sedationi
  Frequency domain results Total power (ms2) Low frequency (ms2) High frequency (ms2) LF/HF ratio

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
If a reasonable personal request exist, the investigators can share the data personally.